CLINICAL TRIAL: NCT01082640
Title: A Multicenter, Randomized, Double-Blind, Phase 2 Study to Evaluate the Effect of Febuxostat Versus Placebo on Renal Function in Gout Subjects With Hyperuricemia and Moderate to Severe Renal Impairment
Brief Title: Effect of Febuxostat on Renal Function in Patients With Gout and Moderate to Severe Renal Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMX-67_203; U1111-1113-8008 (Registry Identifier: WHO)
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Renal Impairment
Keywords: Gout; physiology; Hyperuricemia; Uric Acid; Drug Therapy
MeSH Terms: conditions — Renal Insufficiency; Gout; Hyperuricemia | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo-matching capsules, orally, twice daily for up to 12 months.
  Interventions: Drug: Placebo
- Febuxostat 30 mg BID (Experimental): Febuxostat 30 mg, capsules, orally, twice daily (BID) for up to 12 months.
  Interventions: Drug: Febuxostat
- Febuxostat 40/80 mg QD (Experimental): Participants initially received febuxostat 40 mg, capsules, once daily (QD) and one placebo-matching capsule QD and remained on this dose for up to 12 months if their serum urate (sUA) was <6.0 mg/dL at the Day 14 visit. Participants whose sUA was ≥6.0 mg/dL at the Day 14 visit received febuxostat 80 mg, capsule, QD, and one placebo-matching capsule QD at the Month 1 visit, and for the remainder of the study.
  Interventions: Drug: Febuxostat; Drug: Placebo

INTERVENTIONS:
Drug: Febuxostat — Febuxostat capsules
  Other Names: Uloric; TMX-67
  Arms: Febuxostat 30 mg BID; Febuxostat 40/80 mg QD
Drug: Placebo — Febuxostat placebo-matching capsules
  Arms: Febuxostat 40/80 mg QD; Placebo

SUMMARY:
The purpose of this study is to determine the effect of febuxostat, once daily (QD) or twice daily (BID), on renal function in gout patients with elevated serum urate levels and who have moderate to severe renal impairment.

DETAILED DESCRIPTION:
Gout is caused by high levels of uric acid in the body, and is associated with a broad range of conditions including heart disease, chronic kidney disease and high blood pressure. Hyperuricemia, which is defined as an elevation in serum urate levels, develops into gout when urate crystals form in the body and settle in joints and other organs.

Approximately 40-60% of patients with hyperuricemia and gout have some degree of renal impairment. Hyperuricemia has long been associated with renal disease, and chronic hyperuricemia as seen in gout can lead to deposition of urate crystals resulting in diminished renal function.

This study will evaluate the effect of febuxostat on the renal function of patients with hyperuricemia and gout and moderate to severe renal impairment.

All participants must have an average sitting blood pressure measurement less than 160 mmHg systolic and less than 95 mmHg diastolic. All participants must meet the American Rheumatism Association (ARA) diagnostic criteria for gout (subjects with tophi were excluded). Participants are expected to return to the site for approximately 10 visits.

ELIGIBILITY:
Inclusion Criteria:

* Must have a serum urate greater than 7 mg/dL and a serum creatinine greater than or equal to 1.5 mg at Day -21
* Must have a history or presence of gout defined as having one or more of the American Rheumatism Association criteria for the diagnosis of gout (the criteria related to tophi have been excluded for the purpose of the study)
* Must have an estimated Glomerular Filtration Rate (eGFR) of 15 or greater, or less than or equal to 50 mL/min, AND a serum creatinine greater than 1.5 mg/dL at Screening Visit Day -21

Exclusion Criteria:

* Has secondary hyperuricemia (eg, due to myeloproliferative disorder, or organ transplant)
* Has tophaceous gout
* Has a history of xanthinuria
* Has received aspirin greater than 325 mg/day within 35 days prior to Day 1/Randomization Visit
* Has known hypersensitivity or allergy to allopurinol or any component in its formulation
* Has known hypersensitivity to febuxostat or colchicine or any components in their formulation
* Has myocardial infarction or stroke within the 90 days prior to the Screening Visit
* Has alanine aminotransferase and/or aspartate aminotransferase values greater than 2.0 times the upper limit of normal
* Has end stage renal disease or is likely to be a candidate for dialysis over the 1 year study period
* Has a serum creatinine less than or equal to 1.5 mg/dL, or an estimated Glomerular Filtration Rate at Day -21 Screening Visit less than 15 mL/min or greater than 50 mL/min as calculated by the central laboratory
* Is required to take excluded medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (58):
- United States (58):
  - Birmingham, Alabama
  - Peoria, Arizona
  - Sierra Vista, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Huntington Park, California
  - Irvine, California
  - Lakewood, California
  - Long Beach, California
  - Sacramento, California
  - San Diego, California
  - San Jose, California
  - Tustin, California
  - Arvada, Colorado
  - Westminster, Colorado
  - Wheat Ridge, Colorado
  - Middlebury, Connecticut
  - Brandon, Florida
  - Daytona Beach, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Pinellas Park, Florida
  - Port Charlotte, Florida
  - Port Orange, Florida
  - Augusta, Georgia
  - Conyers, Georgia
  - Dunwoody, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Evergreen Park, Illinois
  - Springfield, Illinois
  - Valparaiso, Indiana
  - Wichita, Kansas
  - Elizabethtown, Kentucky
  - Paducah, Kentucky
  - Baltimore, Maryland
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Brooklyn Center, Minnesota
  - Neptune City, New Jersey
  - Morganton, North Carolina
  - Wilmington, North Carolina
  - Fargo, North Dakota
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Bethlehem, Pennsylvania
  - Anderson, South Carolina
  - Greer, South Carolina
  - Chattanooga, Tennessee
  - Houston, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Danville, Virginia
  - Fairfax, Virginia
  - Richmond, Virginia
  - Williamsburg, Virginia
  - Clarksburg, West Virginia
  - Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Saag KG, Whelton A, Becker MA, MacDonald P, Hunt B, Gunawardhana L. Impact of Febuxostat on Renal Function in Gout Patients With Moderate-to-Severe Renal Impairment. Arthritis Rheumatol. 2016 Aug;68(8):2035-43. doi: 10.1002/art.39654. PMID 26894653
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 46 investigative sites in the United States from 09 April 2010 to 31 May 2012.
Pre-assignment Details: Participants meeting the American Rheumatism Association (ARA) diagnostic criteria for gout (subjects with tophi were excluded). were randomized to 1 of 3 arms in a 1:1:1 ratio to receive either febuxostat 40 mg/80 mg once daily (QD) or febuxostat 30 mg twice daily (BID) or placebo for up to 12 months.
Groups:
- Febuxostat 40/80 mg QD: Participants initially received 40 mg febuxostat once daily (QD) and remained on 40 mg QD for up to 12 months if their serum urate (sUA) was <6.0 mg/dL at the Day 14 visit. Participants whose sUA was ≥6.0 mg/dL at the Day 14 visit received febuxostat 80 mg QD at the Month 1 visit, and for the remainder of the study.
Period: Overall Study
Arm/Group | Placebo | Febuxostat 30 mg BID | Febuxostat 40/80 mg QD
Started | 32 | 32 | 32
Completed | 15 | 17 | 24
Not Completed | 17 | 15 | 8
Not completed — Adverse Event | 9 | 5 | 3
Not completed — Withdrawal by Subject | 3 | 3 | 2
Not completed — Major protocol deviation | 3 | 3 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Other | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Febuxostat 30 mg BID | Febuxostat 40/80 mg QD | Total
Number analyzed (Participants) | 32 | 32 | 32 | 96
Age Continuous [Mean (Standard Deviation); unit: years] | 66.3 (12.05) | 67.3 (11.11) | 63.6 (8.15) | 65.7 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 6 | 19
  Male | 26 | 25 | 26 | 77
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3 | 2 | 3 | 8
  Not Hispanic or Latino | 29 | 30 | 29 | 88
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 1 | 3
  Black or African American | 4 | 5 | 7 | 16
  White | 25 | 24 | 21 | 70
  Other | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 32 | 96
Height [Mean (Standard Deviation); unit: cm] | 172.6 (11.55) | 173.8 (9.60) | 172.8 (9.48) | 173.1 (10.16)
Weight [Mean (Standard Deviation); unit: kg] | 100.7 (27.54) | 98.8 (19.84) | 102.6 (25.85) | 100.7 (24.42)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.3 (6.36) | 32.8 (6.45) | 34.2 (7.30) | 33.4 (6.67)
Prior Use of ARB or ACEi [Number; unit: participants] — ARB = angiotensin receptor blocker ACEi = angiotensin converting enzyme inhibitors
  participants
    Angiotensin receptor blocker (ARB) | 8 | 8 | 8 | 24
    Angiotensin converting enzyme inhibitors (ACEi) | 13 | 13 | 13 | 39
    None | 11 | 11 | 11 | 33
Renal History Based on Creatinine Clearance [Number; unit: participants] — Estimated creatinine clearance based on estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease (MDRD) calculation. Moderately impaired = eGFR ≥ 30-50 mL/min, Severely impaired = eGFR ≥ 15- 29 mL/min.
  participants
    Severely impaired | 17 | 9 | 10 | 36
    Moderately impaired | 15 | 23 | 22 | 60
Serum creatinine level [Number; unit: participants]
  Less than 2.0 mg/dL | 10 | 13 | 14 | 37
  2.0 to <2.5 mg/dL | 7 | 13 | 9 | 29
  Greater than 2.5 mg/dL | 15 | 6 | 9 | 30
Serum Urate [Mean (Standard Deviation); unit: mg/dL] | 10.8 (1.96) | 10.4 (1.43) | 10.4 (1.70) | 10.5 (1.70)
Serum Urate Categories [Number; unit: participants]
  <9.0 mg/dL | 7 | 5 | 4 | 16
  9.0 to <10.0 mg/dL | 6 | 6 | 10 | 22
  ≥10 mg/dL | 19 | 21 | 18 | 58
Gout flares in the past year [Number; unit: participnts] — Not all participants had a gout flare within the last year.
  participnts
    1-3 flares | 21 | 16 | 19 | 56
    4-6 flares | 4 | 8 | 3 | 15
    More than 6 | 2 | 3 | 5 | 10
Time since last gout flare [Number; unit: participants]
  Less than 1 month ago | 5 | 5 | 5 | 15
  1 to less than 4 months ago | 2 | 7 | 5 | 14
  4 to less than 6 months ago | 4 | 4 | 2 | 10
  6 to less than 12 months ago | 14 | 8 | 11 | 33
  more than 1 year ago | 7 | 8 | 9 | 24
Previous urate-lowering therapy [Number; unit: participants] — Participants may have received more than one urate-lowering therapy.
  participants
    Febuxostat | 0 | 5 | 2 | 7
    Allopurinol | 19 | 22 | 21 | 62
    Probenecid | 0 | 0 | 1 | 1
    None | 11 | 6 | 9 | 26
    Other | 3 | 2 | 2 | 7
Number of Lifetime Kidney Stone Episodes [Mean (Standard Deviation); unit: episodes] | 4.8 (3.90) | 3.0 (1.67) | 1.8 (1.78) | 2.8 (2.56)
Kidney Stone Passage [Number; unit: participants] — The number of participants with kidney stone episodes was 5, 6 and 11 in each treatment arm respectively.
  participants | 2 | 1 | 3 | 6
Composition of most recent passed stone [Number; unit: participants] — Number of participants with a kidney stone passage was 2, 1 and 3 in each treatment arm respectively.
  participants
    Calcium Oxalate | 1 | 0 | 1 | 2
    Uric acid | 1 | 0 | 1 | 2
    Calcium citrate | 0 | 0 | 1 | 1
    Mixed | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 12 in Serum Creatinine
Description: Renal function was assessed by measuring the change from Baseline in serum creatinine. Analyses were conducted by the Central Laboratory.
Time Frame: Baseline and Month 12
Population: Full analysis set, including all patients who were randomized and received at least 1 dose of double-blind study medication. Only patients with both a baseline value and at least 1 value during the double-blind treatment period are included in the analysis. Missing data were imputed as carrying forward the last observed post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Febuxostat 30 mg BID | Febuxostat 40/80 mg QD
Number analyzed (Participants) | 32 | 32 | 31
mg/dL
  Baseline | 2.52 (0.126) | 2.10 (0.126) | 2.22 (0.128)
  Change from Baseline at Month 12 | 0.19 (0.094) | 0.09 (0.093) | 0.23 (0.094)
Statistical Analysis 1: Comparison: Placebo vs Febuxostat 30 mg BID; All statistical tests were two sided and conducted at the 0.05 significance level; Test type: Superiority or Other; p = 0.459, ANCOVA — No adjustment for multiplicity was made; The model included treatment as a factor, and the baseline value and prior use of an ARB or an ACEi or none as covariates; LS mean difference = -0.10, 95% CI 2-sided [-0.37 to 0.17], Standard Error of Mean 0.134
Statistical Analysis 2: Comparison: Placebo vs Febuxostat 40/80 mg QD; All statistical tests were two sided and conducted at the 0.05 significance level; Test type: Superiority or Other; p = 0.789, ANCOVA — No adjustment for multiplicity was made; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.04, 95% CI 2-sided [-0.23 to 0.30], Standard Error of Mean 0.133

2. Secondary Outcome: Change From Baseline to Month 12 in Estimated Glomerular Filtration Rate (eGFR)
Description: Change from baseline to Month 12 in estimated Glomerular Filtration Rate (eGFR) using the Modification of Diet in Renal Disease (MDRD) formula (as calculated by the central laboratory).
Time Frame: Baseline and Month 12
Population: Full analysis set with available data at Baseline. and at least 1 post-baseline value. Missing data was imputed as carrying forward the last post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m²
Arm/Group | Placebo | Febuxostat 30 mg BID | Febuxostat 40/80 mg QD
Number analyzed (Participants) | 32 | 32 | 31
mL/min/1.73m²
  Baseline | 29.31 (1.461) | 34.14 (1.461) | 34.08 (1.484)
  Change from Baseline at Month 12 | -2.05 (1.198) | 0.33 (1.172) | -0.86 (0.190)
Statistical Analysis 1: Comparison: Placebo vs Febuxostat 30 mg BID; Test type: Superiority or Other; p = 0.162, ANCOVA — No adjustment for multiplicity was made; [statistical method as in outcome 1, analysis 1]; LS mean difference = 2.38, 95% CI 2-sided [-0.97 to 5.73], Standard Error of Mean 1.687
Statistical Analysis 2: Comparison: Placebo vs Febuxostat 40/80 mg QD; Test type: Superiority or Other; p = 0.485, ANCOVA — No adjustment for multiplicity was made; [statistical method as in outcome 1, analysis 1]; LS mean difference = 1.19, 95% CI 2-sided [-2.18 to 4.57], Standard Error of Mean 1.698

3. Secondary Outcome: Percentage of Participants With Serum Urate (sUA) Less Than 6 mg/dL at Month 12
Description: Serum urate concentrations were determined using the enzymatic method as performed by the Central Laboratory.
Time Frame: Month 12
Population: Full analysis set, including all patients who were randomized and received at least 1 dose of double-blind study medication. A patient was included in the analysis only when there was at least 1 value during the double-blind treatment period. Missing data were imputed as carrying forward the last observed post-baseline value.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Febuxostat 30 mg BID | Febuxostat 40/80 mg QD
Number analyzed (Participants) | 32 | 32 | 31
percentage of participants | 0 | 68.8 | 45.2
Statistical Analysis 1: Comparison: Placebo vs Febuxostat 30 mg BID; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Prior use of an ARB, ACEi, or none was a stratification variable
Statistical Analysis 2: Comparison: Placebo vs Febuxostat 40/80 mg QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Prior use of an ARB, ACEi, or none was a stratification variable
Statistical Analysis 3: Comparison: Febuxostat 30 mg BID vs Febuxostat 40/80 mg QD; Test type: Superiority or Other; p = 0.062, Cochran-Mantel-Haenszel; Prior use of an ARB, ACEi, or none was a stratification variable

4. Secondary Outcome: Mean Clearance (CL/F) of Febuxostat at Steady State
Description: Mean CL/F at steady state were estimated using a population pharmacokinetic (PK) approach, based on 2 PK samples collected prior to dosing, and 4 PK samples collected postdose.
Time Frame: The 2 pre-dose PK samples collected were collected at any 2 of the following visits: Months 3, 6, 9, and/or 12, at -0.25 to 0 hours. The 4 postdose PK samples were collected at Months 3, 6, and/or 9, at 0.25; 0.75 to 2.0; 2.5 to 4.0; and 5 to 12 hours.
Population: Participants who received febuxostat and had available data for PK analysis.
Measure: Mean (Standard Deviation); unit: liters/hour
Groups:
- Febuxostat 40 mg QD: Participants initially received 40 mg febuxostat once daily (QD) and remained on 40 mg QD for up to 12 months if their serum urate (sUA) was <6.0 mg/dL at the Day 14 visit.
- Febuxostat 80 mg QD: Participants with serum urate levels ≥6.0 mg/dL at the Day 14 visit received febuxostat 80 mg QD from the Month 1 visit through Month 12.
Arm/Group | Febuxostat 30 mg BID | Febuxostat 40 mg QD | Febuxostat 80 mg QD
Number analyzed (Participants) | 25 | 9 | 20
liters/hour | 8.16 (2.31) | 8.71 (2.21) | 10.9 (4.70)

5. Secondary Outcome: Mean Area Under the Concentration-Time Curve During the Dosing Interval (AUC[0-τ]) of Febuxostat at Steady State
Description: Mean AUC during the dosing interval at steady state was estimated using a population pharmacokinetic (PK) approach, based on 2 PK samples collected prior to dosing, and 4 PK samples collected postdose.
Time Frame: as for outcome 4
Population: Participants who received febuxostat and had available data for PK analysis.
Measure: Mean (Standard Deviation); unit: hr*µg/mL
Arm/Group | Febuxostat 30 mg BID | Febuxostat 40 mg QD | Febuxostat 80 mg QD
Number analyzed (Participants) | 25 | 9 | 20
hr*µg/mL | 3.98 (1.21) | 4.91 (1.29) | 8.21 (2.30)

ADVERSE EVENTS:
Time Frame: From first double-blind dose date and up to 30 days after the last dose.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Febuxostat 30 mg BID | Febuxostat 40/80 mg QD
Serious Adverse Events (participants affected / at risk) | 7/32 | 5/32 | 8/32
Other Adverse Events (participants affected / at risk) | 20/32 | 21/32 | 23/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | Febuxostat 30 mg BID (N=32) | Febuxostat 40/80 mg QD (N=32)
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 1
Cardiogenic Shock (Cardiac disorders) | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 2 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 2
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Adverse Drug Reaction (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 2 | 1 | 1
Renal Failure Chronic (Renal and urinary disorders) | 0 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
Iliac Artery Occlusion (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | Febuxostat 30 mg BID (N=32) | Febuxostat 40/80 mg QD (N=32)
Blood creatinine increased (Investigations) | 1 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3
Renal impairment (Renal and urinary disorders) | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 4
Nausea (Gastrointestinal disorders) | 3 | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3
Hepatic enzyme increased (Investigations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 2 | 3 | 0
Oedema peripheral (General disorders) | 2 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1
Hypotension (Vascular disorders) | 0 | 0 | 3
Drug hypersensitivity (Immune system disorders) | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 1 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
C-Reactive protein increased (Investigations) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 1
Hypertension (Vascular disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.